CLINICAL TRIAL: NCT01596881
Title: Using OCT to Capture Retinal Microvascular Changes Associated With MS
Brief Title: Using Optical Coherence Tomography to Capture Retinal Microvascular Changes Associated With Multiple Sclerosis
Acronym: OCT in MS
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Rebecca Spain, MD, MSPH, Assistant Professor of Neurology, Oregon Health and Science University
Other Study IDs: OHSU IRB #00008179-MS
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Blood flow; Optical Coherence Tomography; Imaging
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Multiple Sclerosis Patients: Physician-confirmed diagnosis of multiple sclerosis. Any subtype is acceptable. For example, relapsing-remitting, secondary progressive, primary progressive
- Healthy Normal Subjects: Volunteers with healthy eyes.

SUMMARY:
Recent studies have shown that people with multiple sclerosis (MS) who also have diseases related to vascular health such as high cholesterol, high blood pressure, diabetes, cardiovascular disease, and others, may end up more disabled than people with MS who don't have those diseases. This has led to a growing interest in the role of vascular diseases in MS since they may provide another avenue of MS treatment. Some also think that vascular disease may even be a cause of MS. The back of the eye, the retina, is well-suited to studying vascular diseases as blood vessels can be seen even on routine examination of the eye by eye doctors. These specialists are used to seeing changes in retinal blood vessels due to diseases known to affect the eyes such as glaucoma and diabetes. Sophisticated techniques for examining the retina allow for not only visualization of blood vessels, but the rate of blood flow through the blood vessels as well. These blood flow changes are thought to come before changes in what the blood vessels look like, and so may be able to detect problems even earlier than routine examination of the retina by eye doctors. Retinal blood flow has never been carefully studied in MS. Given that MS affects the retina due to the late effects of inflammation of the optic nerve, or optic neuritis, the investigators expect to see altered blood flow in the retinal blood vessels of people with MS compared to healthy control subjects. If so, the investigators can then use retinal blood flow as a way to measure therapies that target vascular diseases in the MS population and determine if those therapies can alter the course of disease.

DETAILED DESCRIPTION:
Background data including age, sex, medical history, and neurologic history and status will be gathered prior to the study/OCT testing visit. At the single study/testing visit, subjects will have their blood pressure and intraocular pressure checked (using numbing drops that last 15-20 minutes), undergo vision testing and then have their eyes dilated with standard dilating drops. They will then undergo optical coherence tomography testing to determine the blood flow of the retinal blood vessels and to take other measurements of the back of the eye including thicknesses of the nervous tissue elements of the retina.

OCT Procedure: The subject will be seated and have their head positioned on a chin rest. They will be asked to look at a target (a lighted spot) while a beam of light scans the front part of the eye. The light is infrared and will not be visible or cause any sensation. A cotton tip swab may be used to help hold the eyelid open temporarily if necessary.

ELIGIBILITY:
Inclusion Criteria (Subjects with MS):

* Physician-confirmed diagnosis of MS (any subtype acceptable, e.g. relapsing- remitting, secondary progressive, primary progressive)
* Age 18-70 years old
* Able to comply with study procedures
* Corrected visual acuity at least 20/200 in either eye

Inclusion Criteria (Healthy subjects):

* Age 18-70 years old
* Able to comply with study procedures
* Able to maintain stable fixation for OCT imaging
* Corrected visual acuity of at least 20/40 in either eye

Exclusion Criteria (all participants):

* Intravenous or oral steroids in the prior 30 days
* Evidence on ophthalmological exam within the last year of other ocular diseases or pathology that would confound the assessment of MS and optic nerve head (e.g. glaucoma, diabetic or hypertensive retinal disease, amblyopia, etc.)
* Previous intraocular surgery except for uncomplicated cataract surgery
* Inability to maintain stable fixation for OCT imaging
* Refractive error greater than +3 or -7 diopters
* MS exacerbation in the prior 60 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll both males and females and include all ethnic and racial groups through clinical practices. The study will enroll subjects from 18 to 70 years of age. Participants older than 70 years are excluded as cooperation with tests may be difficult. For similar reasons, participants who have MS and vision worse than 20/200 are excluded. The study also excludes those with any eye disease that would interfere with of assessment of MS. Otherwise people with any health status are eligible for enrollment. Two groups of participants are recruited: people with healthy, normal eyes and people with any type of MS.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-04; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with MS who also have reduced blood flow in the retina and/or changes in the blood flow to the retina compared to healthy subjects | 1 year

SECONDARY OUTCOMES:
Number of patients with MS who have different blood flow response than healthy subjects to visually stimulating patterns. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spain, MD, MSPH, Principal Investigator — Oregon Health & Science Universtiy
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States